CLINICAL TRIAL: NCT04480983
Title: Role of Multidetector Computerized Tomography (MDCT) in Diagnosis of Non Traumatic Acute Abdomen in Pediatric Age Group.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amal Fathy Abo Elgarad (Other)
Responsible Party: Sponsor-Investigator, Amal Fathy Abo Elgarad, doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: MDCT in acute abdomen
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Acute Abdomen in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Multidetector Computerized Tomography (MDCT) — To evaluate the role of MDCT in diagnosis of non traumatic causes of acute abdomen in pediatric patients with clinical and surgical correlation.

SUMMARY:
To evaluate the role of MDCT in diagnosis of non traumatic causes of acute abdomen in pediatric patients with clinical and surgical correlation.

DETAILED DESCRIPTION:
Acute abdominal pain is a common presenting symptom to the pediatric emergency department (1). The causes of the acute abdomen in pediatric patients are numerous, and diagnosis is often delayed due to misleading signs and symptoms.

Conditions that can be manifested by acute abdominal pain vary in incidence with age and sex. Classification of acute abdominal pain based on age is one adapted approach to narrow the differential diagnosis, which can guide selection of appropriate diagnostic tests, imaging, and definitive treatment.

While most of the emergency visits presenting with acute abdominal pain are self-limited and benign medical diagnoses, a surgical etiology may be present in up to 20%.(7) In nontraumatic cases of an acute abdomen below 1 year of age, the most common surgical etiology was reported to be incarcerated inguinal hernia (45.1%), followed by intussusception (41.9%). These etiologies were uncommon in school-age and adolescent children. In children above 1 year of age, the most common causes of acute surgical diagnoses have been reported to be acute appendicitis , incarcerated hernia, intussusception, intestinal obstruction, and ovarian torsion.

CT scanning provides very detailed images of many types of tissue as well as the lungs, bones, and blood vessels.CT scanning is painless, non invasive and accurate. CT has been shown to be a cost-effective imaging tool for a wide range of clinical problems. CT is less sensitive to patient movement than MRI.

The use of pediatric CT, which is a valuable imaging tool, has been increasing rapidly. However, because of the potential for increased radiation exposure to children undergoing these scans, pediatric CT is a public health concern CT can be a life saving tool for diagnosing illness and injury in children. For an individual child, the risks of CT are small and the individual risk-benefit balance favors the benefit when used appropriately.

Despite the many benefits of CT, a disadvantage is the inevitable radiation exposure.

Radiologists should continually think about reducing exposure as low as reasonably achievable by using exposure settings customized for children. (8,9) There has been revolutionary development in multidetector CT (MDCT) technology that has contributed to a substantial increase in its diagnostic applications and accuracy, even in children. However, a major drawback of MDCT is the use of ionizing radiation and, consequently, the risks of radiation-induced side effects.

It is generally believed that there is a linear-no threshold risk relationship. We should act as if low-dose radiation may well cause secondary cancer and reduce the medical radiation exposure to children as much as possible, the "as low as reasonably achievable" (ALARA) concept.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented by acute abdominal pain from first day of life till fifteen years old.

Exclusion Criteria:

* Patients above 15 years old.
* Patients with traumatic cause of acute abdominal pain.

Ages: 1 Day to 15 Years | Sex: All
Age Groups: Child
Study Population: The role of MDCT in diagnosis of non traumatic causes of acute abdomen in pediatric patients with clinical and surgical correlation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
the role of ultrasound for diagnosis of acute abdominal pain in pediatric. | Baseline
  To evaluate the clinical examination and the role of ultrasound as a primary tool for diagnosis of non traumatic acute abdominal pain in pediatric.

SECONDARY OUTCOMES:
the multidetector CT. | Baseline
  Confirmation of the findings achieved by the primary tools by using the multidetector CT.

REFERENCES:
- [Result] Nievelstein RA, van Dam IM, van der Molen AJ. Multidetector CT in children: current concepts and dose reduction strategies. Pediatr Radiol. 2010 Aug;40(8):1324-44. doi: 10.1007/s00247-010-1714-7. Epub 2010 Jun 10. PMID 20535463